CLINICAL TRIAL: NCT03906721
Title: Reduction of Opioid Dose Using Conditioning & Open-Label Placebo (COLP) in Patients With Spinal Cord Injury, Polytrauma and Burn Injury: A Pilot Study
Brief Title: Reduction of Opioid Dose Using Conditioning & Open-Label Placebo (COLP) in Patients With Spinal Cord Injury, Polytrauma and Burn Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Ross D. Zafonte, MD, Chair, Physical Medicine and Rehabilitation, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001673
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries; Polytrauma; Burn Injury
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Trauma; Burns | interventions — Oxycodone; Oils, Volatile

STUDY DESIGN:
Intervention Model Description: This is a randomized single-blind open-label placebo clinical trial. 60 inpatients will be included from SRH, both men and women aged 18 or older with traumatic and non-traumatic SCI (ASIA A-D), polytrauma and burn injury patients from the Comprehensive Rehabilitation Program at Spaulding Rehabilitation Hospital who have; above, at, or sub-lesional neuropathic pain and/or nociceptive pain (musculoskeletal or visceral) that is moderate or severe in nature (average VAS scale score of 4 or greater at time of enrollment). All subjects must meet clinical criteria for the use of opioids as a treatment for pain management.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conditioning & Open-Label Placebo (COLP) (Experimental): Days 1 to 3 will include the acquisition phase where oxycodone will be prescribed on a schedule of 3-4 times per day and paired with open-placebo and smelling the essential oil. Days 4 to 6 will be the evoked phase, and patients will receive full oxycodone dosage on alternating days with open placebo and smelling the essential oil.
  Interventions: Drug: Placebo; Drug: Oxycodone; Other: Essential Oil
- Treatment-as-usual (Other): For the duration of the study, days 1 to 6, oxycodone will be prescribed on a schedule of 3-4 times per day.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Placebo — Sugar pill used to condition patients.
  Arms: Conditioning & Open-Label Placebo (COLP)
Drug: Oxycodone — An opioid used for analgesia.
  Other Names: Oxycodone Hydrochloride Tablets
Other: Essential Oil — An aromatic oil used for conditioning.
  Arms: Conditioning & Open-Label Placebo (COLP)

SUMMARY:
The use of conditioning open-label placebo (COLP) will be studied as a dose extension method to lower opioid dosage in patients with spinal cord injury, polytrauma, and burn injury. The goal is to provide the same level of pain relief with a reduced opioid dose to diminish adverse effects as well as the risk of addiction associated with narcotic treatment.

DETAILED DESCRIPTION:
The investigators will conduct an assessor blind controlled clinical trial, participants in the COLP group will be fully informed about the interventions the participants will be allocated for. As this study is designed to be a proof-of-concept, only an authorized member of the study staff will be conducting the assessments. Suppose the subject has been approved to participate by the treating physician. In that case, the co-investigator will discuss the study's details and answer questions both before and during the first study visit.

Study Design and Flow:

This study contains one experimental arm and one control group. The experiment will run in a parallel design, with each subject having six days of participation. Each group will have evaluations before starting the trial (Baseline) and assessments after the six days of study participation. Subjects will be evaluated using the following tools: Morphine Equivalent Dose Conversion (MEDC); Modified Brief Pain Inventory (BPI); Spinal Cord Injury - Quality of Life measurement system (SCI-QOL); and Numerical Opioid Side Effects (NOSE). The investigators will also record medication changes, side effects, and pain levels as measured by the Visual Analog Scale (VAS) daily for each patient.

For this open placebo- opioid dose reduction study. The investigators will enroll a total of 60 subjects with SCI, polytrauma, and burn injury patients from the Comprehensive Rehabilitation Program at Spaulding Rehabilitation Hospital and ongoing neuropathic or nociceptive pain. Experimental treatments will take place at either Spaulding Rehabilitation Hospital (SRH). The investigators will coordinate with the appropriate care outlets to ensure that the study's procedures will not interfere with their standard of care at Spaulding. This includes, but is not limited to: physicians, therapists, and nurses working with the patient. The investigators will schedule inpatients as their clinical schedule allows.

After enrollment, subjects will be randomized to receive COLP treatment or to receive standardized opioid dosage.

Oxycodone Intervention and Rescue Medication:

All patients enrolled in this study will receive oxycodone as primary opioid medication for pain control. The treating physician will prescribe a short-acting form of oxycodone 3-4 times per day. The accepted range dosage for this medication will be from 10 to 50 mg PO per day (Q24H), treating physicians will decide the oxycodone dosage to control pain effectively. The investigators expect patients enrolled in this study to take an average of 30-40 mg of oxycodone per day (Q24H).

If a subject requires rescue medication, it will be determined by clinical staff.

Baseline assessments will be performed by the investigators. Subjects on the COLP group will undergo three consecutive days of opioid conditioning paired with taste and odorous placebos (pill and smell), followed by three days of the evoked response phase, where the active opioid medication will be alternated with full placebo dosages to decrease the therapeutic opioid dose by 50%. Females of childbearing age-eligible to participate in the study will be tested for pregnancy using a serum human chorionic gonadotropin (hCG) test.

The treatment regime and schedule for patients in the COLP group will include a short-acting opioid prescribed on a program of 3-4 times per day. This will be considered the active agent for the pharmaco-conditioning intervention; subjects will have access and receive rescue medication if necessary (PRN). Other forms of analgesics (NSAIDs and combos) will be prescribed under the criteria of treating physicians; if combined agents containing opiates are used, a morphine equivalence calculation will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older with traumatic and non-traumatic SCI (ASIA A-D) polytrauma or burn injury patients from the Comprehensive Rehabilitation Program at Spaulding Rehabilitation Hospital,
* SCI, polytrauma or burn injury patients from the Comprehensive Rehabilitation Program at Spaulding Rehabilitation Hospital and pain of no more 5 years of evolution,
* Patients admitted to the Spaulding Comprehensive Rehabilitation Unit at Spaulding Rehabilitation Hospital,
* Who have; above, at, or sub-lesional neuropathic pain and/or nociceptive pain (musculoskeletal or visceral) that is moderate or severe in nature (average VAS scale score of 4 or greater at time of enrollment),
* Respiratory and hemodynamically stable,
* With current narcotic use for pain control,
* Narcotic usage of no more than 120 mg of morphine equivalent

Exclusion Criteria:

* History of alcohol or drug dependence, as self-reported,
* A history of bipolar disorder or psychosis, as self-reported,
* Any substantial decrease in alertness, language reception, or attention that might interfere with understanding,
* Current usage of narcotic medication with dosage higher than 120 mg of morphine equivalent or 80 mg of a short-acting oxycodone,
* Current use of ventilator,
* Compromised medical status due to uncontrolled pathology such as cancer, heart failure, kidney or liver insufficiency, or any other condition which jeopardises patient's participation to the study
* Pregnancy or breastfeeding. Females in childbearing age who are eligible to participate in the study, will be tested for pregnancy by serum hCG test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Morphine Equivalent Dose Conversion (MEDC) | 6 days
  The opioid morphine equivalent conversion factor is used to standardized opioid usage having as a reference morphine as the main indicator for analgesic potency. For drug utilization, there is a need to present usage data consistently, considering dosing requirements. One method of representing opioid use at the population level is through the application of Defined Daily Doses (DDD), however, this represents a problem partly because opioids require highly individualized dosing and need to be titrated to pain response, rather than having standard therapeutic dose ranges. Oral morphine equivalents are based on the idea that different doses of different opioids may give a similar analgesic effect. Where the doses of two different opioids are considered to give a comparable analgesic effect, they are deemed to be equianalgesic doses.

SECONDARY OUTCOMES:
Modified Brief Pain Inventory (BPI) | Day 1 and Day 6
  The BPI is a short self-assessment questionnaire that provides information on various dimensions of pain including how pain developed, the types of pain a patient experiences, and time of day pain is experienced, as well as current ways of alleviating pain. The BPI also consists of the VAS Pain scale, a simple 10- point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine'') measuring a patient' worst pain and least pain, on average and at present time. The Brief Pain Inventory provides information on the intensity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension).
Spinal Cord Injury - Quality of Life measurement system (SCI-QOL) | Day 1 and Day 6
  This measurement system was developed to address the shortage of relevant and psychometrically sound patient reported outcome measures available for clinical care and research in spinal cord injury (SCI) rehabilitation. For the purpose of this research, the Pain Behavior subdomain will be the primary component of this scale to be used. This 7-item fixed-length scale measures manifestations of pain. These actions or reactions can be verbal or non-verbal and involuntary or deliberate. They include observable displays, and verbal reports of pain. This scale includes a small subset of the Patient-Reported Outcomes Measurement Information System (PROMIS ) Pain Behavior item bank (i = 4) and three new items.
Numerical Opioid Side Effects (NOSE) | Day 1 and Day 6
  Opioid therapy may be associated with adverse effects-which may affect the patient's perception of the overall satisfaction with opioid therapy. The Numerical Opioid Side Effect (NOSE) assessment tool is a simple, rapid, self-administered instrument which has the potential to be utilized in a busy pain clinic setting in efforts to document and longitudinally follow trends of opioid adverse effects.
Electroencephalography | Day 1 and Day 6
  Electroencephalography (EEG) is an electrophysiological monitoring method to record the electrical activity of the brain. Quantitative electroencephalography (qEEG) stands out as a valuable, non-invasive tool because it provides reliable and relevant information about brain functioning during rest, sensory stimulation, and cognitive tasks. Besides, this technique is safe, low-cost, and employs a straightforward methodology, making it an appropriate tool for clinical practice. EEG at rest and during pain processing event-related potentials (ERP's) at the patient's bedside. The EEG and ERP recordings will be processed for analytical purposes by the investigators will explore standard EEG metrics (e.g., spectral analysis, connectivity, source localization). At the same time, ERPs will provide information related to pain and values of valence and arousal.
Near-infrared spectroscopy (NIRS) | Day 1 and Day 6
  NIRS is a spectroscopic method that uses the near-infrared region of the electromagnetic spectrum. This method is based on near-infrared light absorption fluctuations that depend on concentration changes of the chromophores O2Hb and HHb in the tissue under investigation. The investigators will use it to investigate the cerebral metabolism of oxygenated (O2Hb), deoxygenated (HHb), and total hemoglobin (tHb) during pain processing ERP. Changes in tHb, defined as the sum of the changes in O2Hb and HHb, can be used to measure blood volume changes. Functional Near-Infrared Spectroscopy (fNIRS) can provide the equivalent of cortical Blood-oxygen-level-dependent (BOLD) signal, similar to functional magnetic resonance imaging (fMRI).
  By combination qEEG and fNIRS data, the investigators will explore the effects of conditioning from a mechanistic perspective; we expect to find some reliable neurophysiological markers associated with the processing of placebo analgesia at a cortical level.
Metabolomics assessment | Day 1 and Day 6
  Metabolomics is the large-scale study of small molecules, commonly known as metabolites, within cells, biofluids, tissues, or organisms. Collectively, these small molecules and their interactions within a biological system are known as the metabolome. The analysis will focus on pathways associated with cognitive and cellular metabolism, metabolites such as indole-3 propionic acid, tryptophan, serotonin, kynurenine, and tyrosine will be analyzed, seeking for alteration associated with cognition. In contrast, uric acid, xanthine, tyrosine, kynurenine, and tryptophan will provide energetic efficiency information. The investigators will collect samples by pinprick system, and analysis will be done using liquid chromatography (LC) technique and by employing Electrochemical Array Detection (ECA).

CONTACTS AND LOCATIONS:
Overall Officials: Ross D Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No